CLINICAL TRIAL: NCT03961633
Title: Asian Women's Action for Resilience and Empowerment (AWARE) Intervention: Feasibility and Efficacy Trial at Three University Health Services Centers
Brief Title: AWARE Intervention: Feasibility and Efficacy Trial at Three University Health Services Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Hyeouk Hahm, Associate Professor, Chair of Social Research, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4755
Record Dates: First submitted 2019-05-10; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Depression; Anxiety; PTSD; Suicidal Ideation; Substance Use Disorders; Unsafe Sex; Coping Behavior
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Suicidal Ideation; Substance-Related Disorders; Unsafe Sex

STUDY DESIGN:
Intervention Model Description: Participants are assigned to a single intervention ("treatment") group. Intervention at the two sites are not concurrent; the Boston University site intervention takes place in March - May 2018, and the Harvard University site intervention takes place in October - December 2018.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AWARE intervention (Experimental): This arm is the "treatment group", which receives the intervention, and is the only arm in the study. See the "intervention" column for more descriptions.
  Interventions: Behavioral: AWARE intervention

INTERVENTIONS:
Behavioral: AWARE intervention — will attend the AWARE group counseling sessions, which are 90 minutes, once a week, for 8 weeks. Each week's session is focused on a specific theme related to the cultural and gender-specific issues typical among young Asian American women. The sessions are led by staff therapists at either institution. For more info on each session's content, please see the "Study Description - Detailed Description" section.
  Participants will fill out forms that detail their therapeutic goals ("commitments") and any adverse emotional / behavioral events from the past week. Participants will also receive daily text messages that reinforce the group session themes.

SUMMARY:
The goal of this study is to test the efficacy and the feasibility of the Asian Women's Action for Resilience and Empowerment (AWARE) intervention, in the real world setting -- student health service centers at Boston University, Wellesley College, and Harvard University.

AWARE is an 8-week group intervention specifically designed to address mental health and sexual health issues among Asian-Pacific Islander (API) women. One AWARE group (final number of 8-10 API women who will be treated) will be held at BU Student Health Services, two groups at Wellesley College, and two groups at Harvard University Health Services for undergraduate and graduate students who meet the demographic and clinical criteria.

During the intervention period, participants will attend the AWARE group counseling sessions, which are 90 minutes, once a week, for 8 weeks. Each week's session is focused on a specific theme related to the cultural and gender-specific issues typical among young Asian American women. The sessions are led by staff therapists at either institution. Participants will fill out forms that detail their therapeutic goals ("commitments") and any adverse emotional/behavioral events from the past week. Participants will also receive daily text messages that reinforce the group session themes.

Participants will be assessed pre- and post-intervention on clinical outcomes, including depression, anxiety, PTSD, and suicidality, using standardized quantitative instruments. This serves to evaluate the efficacy of AWARE at improving mental health outcomes. Participants will also participate in a post-intervention focus group session to evaluate the program's implementation and suggest ways for future improvement.

DETAILED DESCRIPTION:
After institutional review application is approved, study recruitment will begin immediately. Electronic and hard-copy fliers will be disseminated around campus. Fliers will be emailed to Offices of Student Affairs, as well as Asian American student groups, at Boston University and Harvard University. Publicity at Wellesley College will be conducted through the Office of the Dean of Students, Intercultural Education Program. The research group social media (AWSHIP Facebook, Instagram, Twitter, monthly newsletter) will also be used to recruit potential participants. Those who are interested in participating in AWARE will be directed to the AWSHIP website, where the link for the <3 minute demographic survey will be available. The survey will have 6 initial screening question and participants must answer in the affirmative to be eligible for the next recruitment step:

"1. How or where did you hear about our study? Why did our advertisement grab your attention/our outreach effort interest you? 2. Do you self-identify as an Asian American female? 3. What is your marital status? 4. What is your age as of this screening? 5. What languages are you fluent in reading, writing, and speaking? 6. Do you currently have a mobile phone (either a regular phone or a smart phone) with a text-messaging plan?"

Individuals who provide answers that meet the preliminary criteria will receive more detailed information about the study (either by phone or email) within a week. They will be invited to meet with the site coordinator/research assistant to complete the consent form. After participants sign the consent form, they will be asked to complete the clinical assessment in the same room (BUSSW: Rooms 345 or 340, Wellesley: Stone Center Counseling Service offices, Harvard U: Counseling and Mental Health Services offices) using the study laptops. Since the clinical assessments contain questionnaires that ask for details on history of mental health and suicidality, the research team will debrief with the participants asking them about their feelings, ensuring their safety and referring them to care immediately (if needed).

The following questions will be asked in the debrief:

"1. How do you feel after completing the measures? 2. Do you feel safe going about your day? 3. Do you need to talk to someone?"

Once the participant completes the assessment and leaves the room, research coordinators will calculate the scores and inform the PI to help determine if participants meet the threshold criteria based on the results of the clinical screening. The PI will only use the screening questionnaire scored to determine study eligibility. This will be done within 24 hours after the clinical assessment. The research coordinators will contact the participant within 48 hours after the clinical assessment to inform whether they are eligible for the intervention. Eligible participants will be invited to join the intervention group until all the spots have been filled.

The screening questionnaire will contain the following measures:

1. The Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) is a survey that screens for depression by measuring the severity of symptoms linked with depressive episodes. Eligibility criteria is a score equal to or greater than 16.
2. The Hospital Anxiety and Depression Scale (HADS) determines the levels of depression and anxiety that a participant may be experiencing. Eligibility criteria is a score equal to or greater than 11.
3. The PTSD Checklist - Civilian Version (PCL-C) screens for the key symptoms of PTSD that applies to any traumatic event that has happened. Eligibility criteria is a score equal to or greater than 30.
4. As well, exposure to physical or sexual violence during childhood is assessed using the Adverse Childhood Experience International Questionnaire (ACE-IQ). The (ACE-IQ) surveys the first 18 years of the participant's life, such as physical or sexual abuse from household or non-household members.
5. The SF-12 Health Survey (SF-12) asks for personal views on health and keeps track of how the participant feels/how well the participant is able to do perform usual activities.
6. The Columbia-Suicide Severity Rating Scale (C-SSRS) assesses the suicidality of the participant, such as suicidal ideation, intent of ideations, and suicidal behavior. Any participant who indicates that they attempted suicide for the last two years, will be immediately referred to the Student Health Service Center therapist for individual psychotherapy instead of being part of the group intervention.

In addition, for the Harvard University site, the pre-/post-intervention questionnaires will also contain measures that aim to clarify the psychosocial mechanisms through which the AWARE intervention acts to improve mental health outcomes:

1. Frost Multidimensional Perfectionism Scale (MPS) measures the individual's propensity towards perfectionistic thinking and behavior;
2. Distress Tolerance Scale (DTS) measures the individual's capacity and coping behaviors to tolerate emotionally distressful events;
3. Asian American Family Conflict Scale (AAFCS) assesses the conflicts in values and practices between U.S.-raised children and their immigrant parents, in terms of likelihood of occurrence and seriousness of conflict;
4. Multigroup Ethnic Identity Measures (MEIM) assess the individual's commitment (i.e. affirmation and belonging) towards her ethnic identity group, as well as the extent of her exploration and resolution of identity issues;
5. Attitudes Toward Seeking Professional Psychological Help Scale - Short Form (ATSPPHS) measures the participant's stigma toward mental health and seeking psychological help.

Following the screening and consent process, depending on demand, eligible participants may be assigned to a waiting list. Since this is a small study, it is anticipated that some participants may not be able to join the intervention during the clinical trial period. The research team will encourage those who will be unable to join the intervention to participant in any other form of mental health treatment offered at the student health service center. If the participants still want to be part of the intervention, they will be informed that they may be able to participate the following semester.

For Wellesley College, approximately 30 participants are expected to complete the initial demographic screening, and approximately 75% (n = 23) of those women are expected to meet all inclusion criteria on the subsequent clinical screening. Approximately 85% (n = 20) will be both eligible for the inclusion criteria and will commit to 8 weeks of approximately 90 minutes of AWARE intervention.

For Boston University, approximately 30 participants are expected to complete the initial demographic screening, and approximately 75% (n = 23) of those women are expected to meet all inclusion criteria on the subsequent clinical screening. Approximately 40% (n = 10) will be both eligible for the inclusion criteria and will commit to 8 weeks of approximately 90 minutes of AWARE intervention.

For Harvard University, approximately 60 participants are expected to complete the initial demographic screening, and approximately 75% (n= 45) of those women are expected to meet all inclusion criteria on the subsequent clinical screening. Approximately 33% (n= 18-20) will be both eligible for the inclusion criteria and will commit to 8 weeks of approximately 90 minutes AWARE intervention.

The AWARE intervention was developed as a culturally informed treatment that addresses issues of family dynamics, trauma, mental health, and sexual health in Asian American women. The 8 sessions in the AWARE intervention was developed to be sensitive to the gender power dynamics that is consistent throughout many Asian cultures. The sessions provide a safe space for Asian American women to explore the impact of family issues including conflict with parents and family violence as well as understanding coping styles and identity development. The AWARE intervention also addresses mental and physical symptoms that are relevant for trauma survivors. The AWARE intervention was also developed for Asian American women who have experienced Intimate Partner Violence. The sessions focus on how to achieve safety and stability by teaching participants various skills such as how to identify unhealthy relationship patterns and increase safety in their relationships and sexual practices.

Each participant will complete the Adverse Events Log for each week. They will bring the log to each intervention session. The log will take 5-7 minutes to complete. The Adverse Events Log is a form that the subjects will complete to let the therapist know if there were any safety concerns in the previous week.

The topics for the intervention follow the AWARE manual. The topics include:

Session 1: Introduction to AWARE Session 2: "ABCDG" Parenting & Coping with Disempowerment Session 3: Catch-22: The Double Bind Session 4: Who Do I See in the Mirror? Body Image, Stereotypes, & the Media Session 5: Romance, Violence, & Everything in Between Session 6: Sex and Substance Use Session 7: Giving Yourself Grace Session 8: New Beginnings

During the intervention, participants will receive text messages once a day that will provide helpful tips and strategies that promote wellness, encourage self-care, and provide new information and resources. The text messages will not indicate that the subjects are part of a research study.

Examples of text message stories include:

"Being empowered is easier said than done. When you are faced with an emotionally challenging obstacle, you can often act in ways that you feel you are not in control of recognizing your emotions and how you react to them is a key step in discovering how you can empower yourself."

* "STOP is a coping skill that we can use to cope. When we recognize that we are in an emotionally heightened state, take a moment to stop whatever you're doing or thinking, take a deep mindful breath, observe (with your senses and internally), and proceed with caution (respond not react)."
* "More often than not, you are who you are and your perceptions of yourself is connected to your experiences and/or relationship with your parents. Asian-American women often have complicated relationships with their parents; and their actions may confuse you. It is helpful to understand these experiences and this relationship as part of your healing process."

Once the intervention has been completed, the participants will complete the post-test clinical evaluations. These evaluations will be the same as the measures completed during the clinical screening prior to the start of the intervention. The clinical evaluations will be send to the participants after the completion of the final session. The participants will receive an email link with their unique study identification number that they will input when they complete the clinical eligibility screening. The research team will encourage them to complete the clinical screening within 48 hours. This will take about 35-45 minutes.

Participants will be asked to participate in a focus group after the completion of the post-test. The participants are not mandated to take part in the focus group. The focus group will allow the participants to give the principal investigator feedback on the AWARE intervention contents. The focus group discussion will use a semi-structured interview and last approximately 90 minutes.

ELIGIBILITY:
Inclusion Criteria -- participants must meet all of the following:

1. 18 - 35 years old;
2. Identify as Asian American females;
3. Single (unmarried);
4. Have a mobile phone with a text messaging plan;
5. Having depressive symptoms (CESD-R score equal to or greater than 16), or clinical anxiety (HADS-A score equal to or greater than 11), or PTSD symptoms (PCL-C score equal to or greater than 30), or exposure to physical or sexual violence during childhood (assessed using the ACE-IQ).

Exclusion Criteria -- participants who meet any of the following:

1. Actively suicidal and homicidal (assessed using C-SSRS);
2. Participants who show psychotic symptoms such as visual or auditory hallucinations;
3. Students at the trial facilities who are currently members of the research team.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Anyone who self-identifies as an "(Asian American) woman".
Enrollment: 50 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms | Pre/post-intervention (within 4 weeks prior / within 1 week following intervention)
  Change in depression symptoms measured by the Center for Epidemiologic Studies Depression Scale - Revised (CESD-R). The CESD-R scoring scale ranges from 0 (no depression) to 80 (severe depression), and 16 or higher is the threshold for clinical depression diagnosis.
Change in anxiety symptoms | Pre/post-intervention (within 4 weeks prior / within 1 week following intervention)
  Change in depression symptoms measured by the Hospital Anxiety and Depression Scale (HADS). The HADS scoring scale ranges from 0 (no anxiety) to 21 (severe anxiety), and 11 or higher is the threshold for clinical anxiety disorder diagnosis.
Change in PTSD symptoms | Pre/post-intervention (within 4 weeks prior / within 1 week following intervention)
  Change in PTSD symptoms measured by the PTSD Checklist - Civilian Version (PCL-C). The PCL-C scoring scale ranges from 1 (no PTSD symptoms) to 85 (severe PTSD symptoms), and 30 or higher is the threshold for clinical PTSD diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Hyeouk C Hahm, PhD, LCSW, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Boston University Student Health Services, Boston, Massachusetts
  - Harvard University Health Services, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No